CLINICAL TRIAL: NCT03808571
Title: The Association of Cord Blood Nesfatin-1 and Irisin Level With Fetal Doppler Parameters in Pregnancies Complicated With Intrauterine Growth Restricted Fetuses
Brief Title: Cord Blood Nesfatin-1 and Irisin in the Intrauterine Growth Restricted Fetuses
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, erbil karaman, Associate doctor, Yuzuncu Yil University
Other Study IDs: 1
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Nesfatin-1; Irisin; Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cord blood specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Pregnancies complicated with intrauterine growth restricted fetuses
  Interventions: Other: cord blood specimen during the delivery
- Control group: Healthy pregnancies
  Interventions: Other: cord blood specimen during the delivery

INTERVENTIONS:
Other: cord blood specimen during the delivery — The cord blood will be taken during the delivery of baby.

SUMMARY:
: The aim of this study is to investigate Cord blood irisin and nesfatin-1 levels in pregnancies with intrauterine growth retardation and to determine whether they are associated with abnormal fetal doppler findings or not.

DETAILED DESCRIPTION:
This study was conducted at Yüzüncü Yıl University Medical Faculty Obstetrics and Gynecology Clinic. The study group included 34 pregnant women ranged from 18 to 45 years old who have intrauterine growth retardation and underwent ceseraen section. 32 pregnant women who had no abnormality on prenatal follow-up and underwent elective ceserean seciton served as control group. The maternal age, height, weight, body mass index (BMI), systolic and diastolic blood pressures were recorded in both groups of patients. Maternal serum total blood count and biochemical parameters were obtained from the laboratory parameters. Gestational week at birth, birth weight, sex, 1st and 5th minute APGAR scores were recorded. Blood samples were collected from all the cases during the cesarean section for measurmenet of nesfatin-1 and irisin by doubly clamped umbilical cord. Blood samples were immediately centrifuged in sterile tubes and maintained at -80 ° C until assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with intrauterine grwoth rectricted fetuses.
* Healthy pregnancies

Exclusion Criteria:

* Pregnant women with chronic medical conditions
* multiple pregnancies
* fetuses with fetal malfomations or genetic syndromes
* pregnant women older than 45 years old

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
cord blood nesfatn-1 level measurement | 9 months
  cord blood levels of nesfatin-1 in pregnancies with intrauterine growth restricted fetuses and healthy pregnancies.

SECONDARY OUTCOMES:
Cord blood irisin level measurement | 9 months
  ord blood levels of irisin in pregnancies with intrauterine growth restricted fetuses and healthy pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Medical faculty, department of obstetric and gynecology, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided